CLINICAL TRIAL: NCT04747119
Title: The Effect of Muscle Energy Technique on Femoral Meralgia Paraesthesia in Postpartum: A Randomized Controlled Trial
Brief Title: Effect of MET on Meralgia Paraesthesia Postpartum "Muscle Energy Technique"
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/002864
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Meralgia Paresthetica; Femoral Neuropathy
MeSH Terms: conditions — Femoral Neuropathy

STUDY DESIGN:
Intervention Model Description: the control group received the conventional selected exercise program and the study group received the same exercise training program in addition to muscle energy technique
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received the conventional selected exercise program in addition to muscle energy technique
  Interventions: Other: muscle energy technique; Other: conventional selected physical therapy
- control group (Experimental): received the conventional selected exercise program
  Interventions: Other: conventional selected physical therapy

INTERVENTIONS:
Other: muscle energy technique — the patient was supine and the therapist fix the lower limb of the affected side then ask the patient to perform isometric contraction for abductors maintained for 3-5 seconds, then the patient was instructed to stop, exhale and relax then the therapist perform further adducted the patient's knee of the affected side as a stretching exercise for Three to five repetitions of these directions were performed.
  Arms: study group
Other: conventional selected physical therapy — 1. life style modification
  2. Transcutaneous electrical nerve stimulation (TENS)
  3. Flexibility stretching exercises to the hip flexors

SUMMARY:
To investigate the effect of muscle energy technique on Femoral meralgia paraesthesia in a postpartum female. BACKGROUND: meralgia paraesthesia is one of the serious disorders in the postpartum female which results in pain and less physical activities.

………HYPOTHESES:

This study hypothesized that:

muscle energy technique will have a significant effect on Femoral meralgia paraesthesia in postpartum female

DETAILED DESCRIPTION:
Thirty meralgia paraesthesia postpartum females will participate in this study.

The patients will randomly be divided into two equal groups; the control group received the conventional selected exercise program and the study group received the same exercise training program in addition to muscle energy technique, three times per week for four weeks.

The evaluation methods by Femoral nerve conduction velocity will be measured via the Neuropack S1 MEB9004 EMG device before the exercise program and after finishing the exercise program, and also the Pelvic compression test and Pain numeric rating scale

ELIGIBILITY:
Inclusion Criteria:

* Thirty meralgia paraesthesia postpartum female Patients
* with positive Pelvic compression test
* age ranging from 25:40 years
* post vaginal delivery or post-operative (postpartum) persistent dysthesia in anterolateral thigh (one side or both)
* body mass index (20:29.9) Kg/m2

Exclusion Criteria:

* difficulty to communicate or to understand program instructions
* other conditions that caused pain (for example fibromyalgia and arthritis)
* any psychiatric or cognitive symptoms any other musculoskeletal disorders or neurologic diseases of the lower extremities and spine

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all the patients were postpartum females
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Femoral nerve conduction latency | 4 weeks
  Femoral nerve conduction latency measured via the Neuropack S1 MEB9004 EMG device

SECONDARY OUTCOMES:
Pelvic compression test | four weeks
  the therapist applied a downward compression force to the pelvis and maintained a pressure for 45 seconds. If the patients reported an alleviation of symptoms the test is considered positive
Numeric Pain Rating Scale (NPRS) | four weeks
  it includes 11-point numeric scale ranges from no pain with score of "0" to worst pain imaginable with score of "10"

CONTACTS AND LOCATIONS:
Overall Officials: Lama Saad Mahmoud, PHD, Study Chair — October 6 University
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No